CLINICAL TRIAL: NCT03651986
Title: Diagnostic and Monitoring Significance of Circulating Tumor DNA (ctDNA) Methylation Analysis by Next-Generation Sequencing in Benign and Malignant Pulmonary Nodules
Brief Title: Diagnostic and Monitoring Significance of ctDNA Methylation Analysis by NGS in Benign and Malignant Pulmonary Nodules
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AnchorDx Medical Co., Ltd. (Industry)
Collaborators: Xiangya Hospital of Central South University (Other); West China Hospital (Other); Shanghai Zhongshan Hospital (Other); Shanghai Pulmonary Hospital affiliated to Tongji University (Unknown); First Hospital of China Medical University (Other); Guizhou Provincial People's Hospital (Other); Shanghai Chest Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Qilu Hospital of Shandong University (Other); Inner Mongolia People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Second Hospital of Jilin University (Other); LanZhou University (Other); Peking University Third Hospital (Other); The First People's Hospital of Yunnan (Other); Shantou Affiliated Hospital of Sun Yat-Sen University (Unknown); Ruijin Hospital (Other); Tongji Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Air Force Medicial University (Other); Shenzhen People's Hospital (Other); Henan Provincial People's Hospital (Other); Beijing Chao Yang Hospital (Other); Xiamen Second Hospital (Unknown); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Other Study IDs: AnchorDx LC201801
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Nodules
Keywords: Circulating Tumor DNA (ctDNA); DNA Methylation Analysis; Next-Generation Sequencing (NGS); Low-Dose Computed Tomography (LDCT)
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
  Formalin-fixed paraffin-embedded (FFPE) tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort: This is a prospectively enrolling cohort study and a stratified case-cohort design will be employed to select malignant pulmonary nodules cases and benign pulmonary nodules subjects who will be assayed. All participants will be followed up with chest CT or low-dose computed tomography (LDCT) scans for 2-3 years, and take the diagnostic test, ctDNA methylation analysis by NGS, at each visit.
  Interventions: Diagnostic Test: ctDNA methylation analysis by NGS

INTERVENTIONS:
Diagnostic Test: ctDNA methylation analysis by NGS — A blood-based assay for differentiating benign and malignant pulmonary nodules early using circulating tumor DNA (ctDNA) methylation analysis by next-generation sequencing (NGS)

SUMMARY:
AnchorDx is using circulating tumor DNA (ctDNA) methylation analysis by next-generation sequencing (NGS) to develop a blood-based assay for differentiating benign and malignant pulmonary nodules early. The purpose of this study is to evaluate the diagnostic performance of this assay in patients with pulmonary nodules.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational cohort study and seeks to enroll 10,560 participants with pulmonary nodules smaller than 3 cm in diameter from 21 hospitals in China. All participants will be followed up with chest CT or low-dose computed tomography (LDCT) scans for 2-3 years ( baseline, 3 months, 6 months, 12 months, 24 months and 36 months). Their blood samples, CT or LDCT scans data, and clinical data will be collected at each visit and Formalin-fixed paraffin-embedded (FFPE) tissues will be collected when participants who receive pneumonectomy or percutaneous lung biopsy.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* pulmonary nodules diagnosed by chest CT or low-dose computed tomography (LDCT) scans

  * non-calcified pulmonary nodules with the diameter between 5mm to 30mm
  * including solid nodules, mixed ground-glass opacity nodules and pure ground-glass opacity lung modules
* new cases of pulmonary nodules or diagnosed within 60 days prior to enrollment
* agree to finish the Patient Pulmonary History Questionnaire
* agree to be followed up for 2-3 years
* agree to provide a written informed consent

Exclusion Criteria:

* pregnant or lactating women
* received any pneumonectomy or percutaneous lung biopsy before enrollment
* recipients of blood transfusions within 30 days prior to enrollment
* patients with tumors identified within 2 years prior to enrollment except non-melanoma skin cancer
* fail to understand or provide a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with pulmonary nodules diagnosed by chest CT or low-dose computed tomography (LDCT) scans
Sampling Method: Probability Sample
Enrollment: 10560 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance of the blood-based assay for differentiating benign and malignant pulmonary nodules early using circulating tumor DNA (ctDNA) methylation analysis by next-generation sequencing (NGS) | 3 Years
  The efficacy of the blood-based ctDNA methylation assay comparing with pathologic diagnosis, the gold standard, and CT/LDCT diagnosis, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

SECONDARY OUTCOMES:
The diagnostic and monitoring significance of routine tests integrating with ctDNA methylation analysis by NGS in differentiating benign and malignant pulmonary nodules | 3 Years
  The diagnostic performance of the combination of routine tests and ctDNA methylation analysis by NGS in differentiating benign and malignant pulmonary nodules, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan ZHONG, MD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (23):
- China (23):
  - Department of Respiratory and Critical Care Medicine, Beijing Chaoyang Hospital, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - Department of Respiratory Medicine, West China Hospital of Sichuan University, Chengdu
  - Department of Pulmonary Medicine, The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Department of Respiration and Critical Care Medicine, Guizhou Provincial People's Hospital, Guiyang
  - Department of Pulmonary and Critical Care Medicine, Inner Mongolia Autonomous Region People's Hospital, Hohhot
  - Department of Respiratory, QILU Hospital, Shandong University, Jinan
  - Department of Respiratory Medicine, The First People's Hospital of Yunnan Province, Kunming
  - Department of Gerontal Respiratory Medicine, The Frist Hospital of Lanzhou University, Lanzhou
  - Department of Respiration, The First Affiliated Hospital of Nanchang University, Nanchang
  - Department of Pulmonary & Critical Care Medicine, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Department of Pulmonary Medicine, Shanghai Chest Hospital, Shanghai Jiaotong University, Shanghai
  - Department of Pulmonary Medicine, Zhongshan Hospital, Fudan University, Shanghai
  - Department of Respiratory Medicine, Shanghai Pulmonary Hospital, Tongji University School of Medicine, Shanghai
  - Department of Respiratory Medicine, Shantou Central Hospital, Shantou
  - Department of Respiratory Medicine, The First Hospital of China Medical University, Shenyang
  - Department of Respiratory Medicine, Shenzhen People's Hospital, Shenzhen
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Department of Pulmonary and Critical Care Medicine, The First Affiliated Hospital, Xi'an Jiaotong University, Xi'an
  - Department of Pulmonary Medicine, Xijing Hospital, Air Force Medical University of PLA, Xi'an
  - Department of Cardiothoracic Surgery, The Second Affiliated Hospital of Xiamen Medical College, Xiamen
  - Department of Respiratory Medicine, Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang W, Liu D, Li M, Wang W, Qin Z, Zhang J, Zhang Y, Hu Y, Bao H, Xiang Y, Wang B, Wu J, Sun J, Hu C, Ye X, Zhang X, Xiao W, Yun C, Sun D, Wang W, Chang N, Zhang Y, Zhao J, Zhang X, Xu J, Wu D, Liu X, Guo Y, Zhang Q, Zhang W, Yang L, Li Z, Zhang X, Han B, Tong Z, He J, Qu J, Fan JB, Zhong N. Evaluating the diagnostic accuracy of a ctDNA methylation classifier for incidental lung nodules: protocol for a prospective, observational, and multicenter clinical trial of 10,560 cases. Transl Lung Cancer Res. 2020 Oct;9(5):2016-2026. doi: 10.21037/tlcr-20-701. PMID 33209621